CLINICAL TRIAL: NCT03798587
Title: PNA-mediated Inhibition of the SENP1 Molecular Hub as a Potential Therapeutic Approach for the Suppression of Osteosarcoma Growth and Metastasis (PNA-OS)
Brief Title: Inhibition of SENP1 for the Suppression of OS Growth and Metastasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: PNA-OS
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-01

CONDITIONS: Primary Osteosarcoma of Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Wasted biological material derived from osteosarcoma eradication surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OS patients: Patients with age ≥18 years that were/can be recruited within the IRCCS Istituto Ortopedico Galeazzi BioBanca (ethical committee approval n. 29/INT/2017).
  Patients with age <18 years: will be additionally recruited besides the IRCCS Istituto Ortopedico Galeazzi BioBanca.
  The target group corresponds to patients hospitalized at Istituto Ortopedico Galeazzi, undergoing surgical eradication of primary osteosarcoma.
  Patients will be considered eligible for enrollment in the study if able to sign the consent to the procedure after appropriate information from the reference surgeon or signed by parents or legal guardian after appropriate information from the reference surgeon (if age <18).
  Inclusion Criteria:
  * Indication for primary OS eradication surgery
  * Patients hospitalized in Istituto Ortopedico Galeazzi
  Exclusion criteria:
  -Patients not able to sign the Informed Consent.

SUMMARY:
The aim of this project is to test a new powerful PNA-based SENP1 inhibitor, previously characterized in an in vitro model of OS cell lines.

The most effective PNA, conjugated with a cell-permeable CPP, which is able to inhibit OS cells viability and invasiveness in both normoxia and hypoxia through SENP1-mediated inhibition of HIF1α, ZEB1, and Akt, will be investigated for its ability to penetrate and silence SENP1 expression in ex vivo human OS tissues.

Primary aim:

To determine the ability of PNA-CPP to penetrate into an ex vivo tridimensional tissue of OS, derived from wasted biological material obtained during OS eradication surgery, and to exert its biological function of inhibiting SENP1 within the tissue.

DETAILED DESCRIPTION:
Background:

Osteosarcoma (OS) is the most common type of primary malignant bone tumor in children and adolescents. The overall survival rate is dramatically reduced by the development of metastases, often pulmonary. Solid malignant tumors, such as OS, often develop a hypoxic microenvironment, which contributes to tumor growth, metastasis, treatment failure, and patient mortality. Adaptation to hypoxia, as well as to other environmental conditions, is often associated with modifications in the post-transcriptional regulation of key effectors. Among these, SUMOylation is carried out by small ubiquitin-like modifier (SUMO) proteins and is dynamically reversed (deSUMOylation) by Sentrin/SUMO-specific proteases (SENPs). SENP1, the best characterized SENP, is upregulated in multiple tumors being involved in tumorigenesis and tumor progression. Through deSUMOylation, SENP1 acts as a molecular hub that stabilizes and activates key regulator factors, such as hypoxia-inducible factor 1α (HIF1α), zinc finger E-box binding homeobox 1 (ZEB1), and Akt, responsible for tumor cells adaptation to hypoxic microenvironment, induction of cell proliferation, invasion and migration, and inhibition of apoptosis, thus contributing to tumor progression and metastasis.

HIF1α is the master transcriptional regulator for cellular adaptation and survival under hypoxic conditions, and contributes to enhance the cell metastatic potential. SENP1-mediated HIF1α deSUMOylation prevents HIF1α degradation by proteasome, thus activating the HIF1α signaling pathway. SENP1 is overexpressed in OS cells under hypoxic condition and siRNA-mediated silencing of SENP1 decreases tumor cell viability, promotes cell apoptosis, reduces invasiveness, and inhibits the epithelial-mesenchymal transition (EMT).

ZEB1 is involved in tumorigenesis, progression, invasion and metastases in several tumors (e.g. glioblastoma, prostate, lung, liver, and colorectal). ZEB1 silencing in OS cells leads to a reduced caspase-3 activity, NF-κB and iNOS inhibition, overall reduced cell proliferation and increased apoptosis. SENP1 knockdown in hepatocellular carcinoma (HCC) cells decreases ZEB1 and inhibits EMT].

Akt hyper-activation is essential for the onset and progression of tumors, including OS. In astroglioma cells siRNA-mediated inhibition of SENP1 is associated to Akt hypophosphorylation accompanied by the inhibition of its downstream targets Bcl-xL and cyclinD1 and p21 upregulation, leading to cell-cycle arrest and increased apoptosis.

Altogether, these studies suggest that SENP1 acts as a hub whose inhibition reflects on multiple targets some of which, i.e. HIF1α, ZEB1, Akt, are key factors in tumor progression and metastasis in both normoxia and hypoxia. While it is known the effect of SENP1 on HIF1α in OS, it is reasonable to assume that SENP1 might mediate ZEB1 downregulation and Akt inactivation also in OS. Thus, novel SENP1 inhibition strategies are potentially effective therapeutic approaches to block OS growth and metastasis.

SENP1 inhibition can be achieved by gene silencing mediated by siRNAs. However, naked siRNAs are highly unstable and liposome-based delivery systems are poorly efficient and cytotoxic both in vitro and in vivo. A promising approach for inhibition of SENP1 expression is gene silencing mediated by peptide nucleic acids (PNA), nucleobase oligomers with the phosphate backbone replaced by a pseudopeptide backbone of repeated units of N-(2-aminoethyl) glycine. Because of their unnatural backbone, PNAs are definitively resistant to both nuclease and protease activities, form a more specific and stable binding with the complementary DNA or RNA, allowing an efficient and persistent silencing effect. Although PNA cell permeability is very poor, it can be effectively enhanced by their conjugation with cell-penetrating peptides (CPP). In the last years, PNA have emerged as really promising tools for cancer diagnosis and therapy, and, above all, as effective candidates for stable gene silencing in gene therapy.

Rational and preliminary study:

3 different PNA sequences targeting different SENP1 mRNA regions will be designed and tested. PNAs will be conjugated to an octa-arginine (R8) CPP that efficiently mediate the intracellular delivery of PNAs. The uptake will be studied with a scrambled-sequence R8- and fluorescein (Fl)-conjugated PNA (scrPNA-R8-Fl).

An in vitro characterization of the ability of the designed PNA-CPP to penetrate intracellular and to silence the target SENP1 will be performed in cell lines of OS.

To study the PNA-R8 uptake in OS cells, different OS cell lines (SaOS-2, MG-63, U2OS) with different invasive potential and all expressing SENP1, and primary human osteoblasts (hOb) as negative control for SENP1 expression, will be used. Following incubation with scrPNA-R8-Fl at different concentrations the uptake will be determined at consecutive time-points by flow cytometry, while the cytoplasmic localization will be confirmed by fluorescence microscopy. A scrPNA-Fl not conjugated to R8 will function as a negative control, as it is not expected to enter the cell. Cytotoxicity of scrPNA-R8 will be assayed by Alamar Blue Cell Viability assay. The silencing effectiveness of the different anti-SENP1 PNA-R8 conjugates (senpPNA-R8) will be assayed in all cell lines in both normoxia and hypoxia (1% O2, 5% CO2, and 94% N2). The senpPNA-R8-mediated SENP1 silencing efficiency will be assessed by RT-qPCR and western-blot (WB). scrPNA-R8 will serve as negative control, while cells transfected with siRNA targeting SENP1 will serve as positive control. In this part the most efficient silencing senpPNA-R8 compound will be selected.

The senpPNA-R8-mediated downregulation of HIF1α, and potentially of ZEB1 expression and Akt phosphorylation inhibitions, as consequence of SENP1 inhibition in OS cells, will be assayed by WB. Thus, reduced cell viability, migration and invasion, induction of apoptosis, and EMT inhibition will be assayed, and compared to the effects in hOb. Cell viability will be determined by Alamar Blue assay, whereas apoptosis will be assayed by flow cytometry by staining of Annexin V and with propidium iodide. The residual migration and invasion ability will be assessed by wound-healing assay and transwell invasion assay, respectively. Downregulation of vimentin and N-cadherin and upregulation of E-cadherin, EMT markers and of the downstream targets of ZEB1 (caspase-3, NF-κB) and Akt, (cyclinD1 and Bcl-xL) will be determined by WB.

The in vitro characterization of the penetration and silencing ability of the designed PNA-CPP in OS cell lines is the preliminary step of the study. An ex vivo analysis of the ability of the PNA-CPP to penetrate into a 3D tissue and silence the target SENP in an OS tissue explant from patients will follow.

Aims of the study:

The aim of this project is to test a new powerful PNA-based SENP1 inhibitor, previously characterized in an in vitro model of OS cell lines.

The most effective PNA, conjugated with a cell-permeable CPP, which is able to inhibit OS cells viability and invasiveness in both normoxia and hypoxia through SENP1-mediated inhibition of HIF1α, ZEB1, and Akt, will be investigated for its ability to penetrate and silence SENP1 expression in ex vivo human OS tissues.

Primary aim:

To determine the ability of PNA-CPP to penetrate into an ex vivo tridimensional tissue of OS, derived from wasted biological material obtained during OS eradication surgery, and to exert its biological function of inhibiting SENP1 within the tissue.

Study design:

For this study, wasted biological material derived from osteosarcoma eradication surgery will be collected which comprise only a small proportion of the removed tumor mass other than that used for histological and molecular diagnosis.

15 patients with primary OS will be recruited. The target group will comprise patients hospitalized at IRCCS Istituto Ortopedico Galeazzi who will be subjected to surgical eradication of primary OS.

The study will be presented to patients with age ≥18 years that can be recruited also in the IRCCS Istituto Ortopedico Galeazzi BioBanca protocol (ethical committee approval n. 29/INT/2017) by the surgeon. These patients will sign two Informed Consents: one for the BioBanca and one for the PNA-OS study.

Patients with age <18 years will be additionally recruited besides the IRCCS Istituto Ortopedico Galeazzi BioBanca. These patients will be considered eligible for the study if the legal tutor will sign the Informed Consents relative to the PNA-OS study.

Also samples of OS already existing in the BioBanca as frozen samples preserved in liquid nitrogen at BioRep Service-Provider (BioRep S.r.l. Via Olgettina 60, 20132, Milano), will be used. Every reasonable effort will be done to call these patients to sign a specific informed consent relative to this study.

Since several practical issues (e.g. unsuitableness or low amount of biological material) can occur, we envision the possibility to recruit additional patients until the achievement of 15 complete samples.

The Study will start after approval of Ethical Committee and the estimated duration is 36 months, divided as following:

* Timing for enrolment: 24 month
* Data analysis: 12 month

Experimental design:

Ex vivo analysis of the PNA-R8 silencing ability in osteosarcoma samples. We will investigate whether senpPNA-R8 is able to penetrate into a tridimensional OS tissue and to exert its silencing effect.

15 OS samples will be collected either in the context of the IRCCS Galeazzi BioBanca (ethical committee approval n. 29/INT/2017) or from newly recruited patients, in collaboration with the C.C.O.O.R.R. equip.

Only wasted biological material derived from surgery will be used without any additional harm to the patients other than the surgery itself and the study does not involve any diagnostic aim or genetic profiling of the samples collected.

OS samples, already existing in the BioBanca as frozen samples preserved in liquid nitrogen at BioRep Service-Provider (BioRep S.r.l. Via Olgettina 60, 20132, Milano), will be used to determine the initial expression levels of SENP1 in OS by RT-qPCR. For this, samples will be homogenized, total RNA will be extracted and RT-qPCR will be performed assaying for SENP1 expression levels.

The remaining samples out of 15, freshly collected, will be preserved in physiological solution until usage. The OS samples will be cut in 3 mm3 pieces, placed in a 24-multiwell culture plate, and cultivated ex vivo as organotypic OS cultures in both normoxia and hypoxia-induced microenvironment under orbital rotation [21-23]. Organotypic tumor tissue maintain the complexity of the original tissue with tumor cells being surrounded by their original microenvironment rather than artificial matrices and this system is particularly advantageous for ex vivo drug screening, for studying drug uptake and molecular processes. OS cultures will be treated with senpPNA-R8, and SENP1 expression in naïve and PNA-treated samples will be determined by RT-qPCR and immunohistochemistry in paraffin-embedded sections. The ability of the PNA-R8 to penetrate within the hypoxic core of the OS samples will be assessed: after incubation with scrPNA-R8-Fl, sections will be immediately frozen (-80°C), processed and analyzed by immunofluorescence.

Samples will be analyzed and stored at Laboratorio di Biochimica Sperimentale e Biologia Molecolare at the Istituto Ortopedico Galeazzi for the whole duration of the study. At the end of the study every residual material will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Indication for primary OS eradication surgery
* Patients hospitalized in Istituto Ortopedico Galeazzi

Patients with age ≥18 years: were/can be recruited within the IRCCS Istituto Ortopedico Galeazzi BioBanca (ethical committee approval n. 29/INT/2017).

Patients with age <18 years: will be additionally recruited besides the IRCCS Istituto Ortopedico Galeazzi BioBanca.

Exclusion Criteria:

* Patients not able to sign the Informed Consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 15 patients with primary OS.
  Patients with age ≥18 years that were/can be recruited within the IRCCS Istituto Ortopedico Galeazzi BioBanca (ethical committee approval n. 29/INT/2017).
  Patients with age <18 years: will be additionally recruited besides the IRCCS Istituto Ortopedico Galeazzi BioBanca.
  The target group corresponds to patients hospitalized at Istituto Ortopedico Galeazzi, undergoing surgical eradication of primary osteosarcoma.
  Patients with age ≥18 will be considered eligible for enrollment in the study if able to sign the consent to the procedure after appropriate information from the reference surgeon.
  Patients with age <18 will be considered eligible for enrollment in the study if able to provide the consent to the procedure (donation of waste material) signed by parents or legal guardian after appropriate information from the reference surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Determination of SENP1 expression in OS samples | 8 months
  OS samples, already existing in the BioBanca as frozen samples preserved in liquid nitrogen at BioRep Service-Provider (BioRep S.r.l. Via Olgettina 60, 20132, Milano), will be used to determine the initial expression levels of SENP1 in OS by RT-qPCR. For this, samples will be homogenized, total RNA will be extracted and RT-qPCR will be performed assaying for SENP1 expression levels.
Ex vivo analysis of the PNA-R8 silencing ability in osteosarcoma samples. | 16 months
  Freshly collected OS samples will be preserved in physiological solution until usage. The OS samples will be cut in 3 mm3 pieces, placed in a 24-multiwell culture plate, and cultivated ex vivo as organotypic OS cultures in both normoxia and hypoxia-induced microenvironment under orbital rotation. OS cultures will be treated with senpPNA-R8, and SENP1 expression in naïve and PNA-treated samples will be determined by RT-qPCR and immunohistochemistry in paraffin-embedded sections. The ability of the PNA-R8 to penetrate within the hypoxic core of the OS samples will be assessed: after incubation with scrPNA-R8-Fl, sections will be immediately frozen (-80°C), processed and analyzed by immunofluorescence.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abarrategi A, Tornin J, Martinez-Cruzado L, Hamilton A, Martinez-Campos E, Rodrigo JP, Gonzalez MV, Baldini N, Garcia-Castro J, Rodriguez R. Osteosarcoma: Cells-of-Origin, Cancer Stem Cells, and Targeted Therapies. Stem Cells Int. 2016;2016:3631764. doi: 10.1155/2016/3631764. Epub 2016 Jun 5. PMID 27366153
- [Result] Cao J, Wang Y, Dong R, Lin G, Zhang N, Wang J, Lin N, Gu Y, Ding L, Ying M, He Q, Yang B. Hypoxia-Induced WSB1 Promotes the Metastatic Potential of Osteosarcoma Cells. Cancer Res. 2015 Nov 15;75(22):4839-51. doi: 10.1158/0008-5472.CAN-15-0711. Epub 2015 Sep 30. PMID 26424695
- [Result] Philip B, Ito K, Moreno-Sanchez R, Ralph SJ. HIF expression and the role of hypoxic microenvironments within primary tumours as protective sites driving cancer stem cell renewal and metastatic progression. Carcinogenesis. 2013 Aug;34(8):1699-707. doi: 10.1093/carcin/bgt209. Epub 2013 Jun 5. PMID 23740838
- [Result] Guan G, Zhang Y, Lu Y, Liu L, Shi D, Wen Y, Yang L, Ma Q, Liu T, Zhu X, Qiu X, Zhou Y. The HIF-1alpha/CXCR4 pathway supports hypoxia-induced metastasis of human osteosarcoma cells. Cancer Lett. 2015 Feb 1;357(1):254-264. doi: 10.1016/j.canlet.2014.11.034. Epub 2014 Nov 18. PMID 25444927
- [Result] Bettermann K, Benesch M, Weis S, Haybaeck J. SUMOylation in carcinogenesis. Cancer Lett. 2012 Mar 28;316(2):113-25. doi: 10.1016/j.canlet.2011.10.036. Epub 2011 Nov 2. PMID 22138131
- [Result] Cui CP, Wong CC, Kai AK, Ho DW, Lau EY, Tsui YM, Chan LK, Cheung TT, Chok KS, Chan ACY, Lo RC, Lee JM, Lee TK, Ng IOL. SENP1 promotes hypoxia-induced cancer stemness by HIF-1alpha deSUMOylation and SENP1/HIF-1alpha positive feedback loop. Gut. 2017 Dec;66(12):2149-2159. doi: 10.1136/gutjnl-2016-313264. Epub 2017 Mar 3. PMID 28258134
- [Result] Zhang W, Sun H, Shi X, Wang H, Cui C, Xiao F, Wu C, Guo X, Wang L. SENP1 regulates hepatocyte growth factor-induced migration and epithelial-mesenchymal transition of hepatocellular carcinoma. Tumour Biol. 2016 Jun;37(6):7741-8. doi: 10.1007/s13277-015-4406-y. Epub 2015 Dec 22. PMID 26695141
- [Result] Xia W, Tian H, Cai X, Kong H, Fu W, Xing W, Wang Y, Zou M, Hu Y, Xu D. Inhibition of SUMO-specific protease 1 induces apoptosis of astroglioma cells by regulating NF-kappaB/Akt pathways. Gene. 2016 Dec 31;595(2):175-179. doi: 10.1016/j.gene.2016.09.040. Epub 2016 Sep 28. PMID 27693211
- [Result] Yee Koh M, Spivak-Kroizman TR, Powis G. HIF-1 regulation: not so easy come, easy go. Trends Biochem Sci. 2008 Nov;33(11):526-34. doi: 10.1016/j.tibs.2008.08.002. Epub 2008 Sep 21. PMID 18809331
- [Result] Wang X, Liang X, Liang H, Wang B. SENP1/HIF-1alpha feedback loop modulates hypoxia-induced cell proliferation, invasion, and EMT in human osteosarcoma cells. J Cell Biochem. 2018 Feb;119(2):1819-1826. doi: 10.1002/jcb.26342. Epub 2017 Sep 27. PMID 28796315
- [Result] Shen A, Zhang Y, Yang H, Xu R, Huang G. Overexpression of ZEB1 relates to metastasis and invasion in osteosarcoma. J Surg Oncol. 2012 Jun 15;105(8):830-4. doi: 10.1002/jso.23012. Epub 2011 Dec 27. PMID 22213004
- [Result] Xu XM, Liu W, Cao ZH, Liu MX. Effects of ZEB1 on regulating osteosarcoma cells via NF-kappaB/iNOS. Eur Rev Med Pharmacol Sci. 2017 Mar;21(6):1184-1190. PMID 28387915
- [Result] Li R, Wei J, Jiang C, Liu D, Deng L, Zhang K, Wang P. Akt SUMOylation regulates cell proliferation and tumorigenesis. Cancer Res. 2013 Sep 15;73(18):5742-53. doi: 10.1158/0008-5472.CAN-13-0538. Epub 2013 Jul 24. PMID 23884910
- [Result] Hoyer J, Neundorf I. Peptide vectors for the nonviral delivery of nucleic acids. Acc Chem Res. 2012 Jul 17;45(7):1048-56. doi: 10.1021/ar2002304. Epub 2012 Mar 28. PMID 22455499
- [Result] Wu JC, Meng QC, Ren HM, Wang HT, Wu J, Wang Q. Recent advances in peptide nucleic acid for cancer bionanotechnology. Acta Pharmacol Sin. 2017 Jun;38(6):798-805. doi: 10.1038/aps.2017.33. Epub 2017 Apr 17. PMID 28414202
- [Result] Oh SY, Ju Y, Park H. A highly effective and long-lasting inhibition of miRNAs with PNA-based antisense oligonucleotides. Mol Cells. 2009 Oct 31;28(4):341-5. doi: 10.1007/s10059-009-0134-8. Epub 2009 Sep 30. PMID 19812898
- [Result] McClorey G, Banerjee S. Cell-Penetrating Peptides to Enhance Delivery of Oligonucleotide-Based Therapeutics. Biomedicines. 2018 May 5;6(2):51. doi: 10.3390/biomedicines6020051. PMID 29734750
- [Result] Song C, Liu W, Li J. USP17 is upregulated in osteosarcoma and promotes cell proliferation, metastasis, and epithelial-mesenchymal transition through stabilizing SMAD4. Tumour Biol. 2017 Jul;39(7):1010428317717138. doi: 10.1177/1010428317717138. PMID 28670958
- [Result] Meijer TG, Naipal KA, Jager A, van Gent DC. Ex vivo tumor culture systems for functional drug testing and therapy response prediction. Future Sci OA. 2017 Mar 27;3(2):FSO190. doi: 10.4155/fsoa-2017-0003. eCollection 2017 Jun. PMID 28670477
- [Result] Naipal KA, Verkaik NS, Sanchez H, van Deurzen CH, den Bakker MA, Hoeijmakers JH, Kanaar R, Vreeswijk MP, Jager A, van Gent DC. Tumor slice culture system to assess drug response of primary breast cancer. BMC Cancer. 2016 Feb 9;16:78. doi: 10.1186/s12885-016-2119-2. PMID 26860465
- [Result] Muff R, Botter SM, Husmann K, Tchinda J, Selvam P, Seeli-Maduz F, Fuchs B. Explant culture of sarcoma patients' tissue. Lab Invest. 2016 Jul;96(7):752-62. doi: 10.1038/labinvest.2016.49. Epub 2016 Apr 25. PMID 27111283
- [Result] van der Kuip H, Murdter TE, Sonnenberg M, McClellan M, Gutzeit S, Gerteis A, Simon W, Fritz P, Aulitzky WE. Short term culture of breast cancer tissues to study the activity of the anticancer drug taxol in an intact tumor environment. BMC Cancer. 2006 Apr 7;6:86. doi: 10.1186/1471-2407-6-86. PMID 16603054